CLINICAL TRIAL: NCT03101098
Title: Retroperitoneal Ligation of Uterine Artery in Total Laparoscopic Hysterectomy for Enlarged Uterus: A Randomized Controlled Trial
Brief Title: Retroperitoneal Ligation of Uterine Artery in Total Laparoscopic Hysterectomy for Enlarged Uterus
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB did not approve this study.
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-02-001
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retroperitoneal hysterectomy (Experimental): In subjects allocated to the experimental group, which the uterine vessels were ligated where it originates from the internal iliac artery,
  Interventions: Procedure: Retroperitoneal liagation of uterine artery
- Classical hysterectomy (Active Comparator): The operative technique of classical total laparoscopic hysterectomy (TLH) performed in the control group was comparable to that of retroperitoneal TLH, except for one that coagulation and transection of uterine artery was achieved using an energy device alongside the cervix
  Interventions: Procedure: Classical ligation of uterine artery

INTERVENTIONS:
Procedure: Retroperitoneal liagation of uterine artery — the site of ligation of uterine artery is the area that it originates from the internal iliac artery during TLH
  Arms: Retroperitoneal hysterectomy
Procedure: Classical ligation of uterine artery — the site of ligation of uterine artery is the area alongside the cervix
  Arms: Classical hysterectomy

SUMMARY:
This randomized trial is aimed to investigate the role of retroperitoneal TLH in enlarge uterus.

DETAILED DESCRIPTION:
Laparoscopic hysterectomy is one of the most common gynecologic surgeries worldwide. Generally, in total laparoscopic hysterectomy (TLH), uterine arteries are coagulated or transected close to the uterus, alongside the cervix, like surgical technique of a conventional total abdominal hysterectomy. Recently, several studies showed that ligation of uterine artery where it originates from the internal iliac artery during TLH (so-called "retroperitoneal TLH") is effective for reducing blood loss. However, the application of this technique to clinical practice have not been well investigated in terms of its efficacy and safety. Moreover, most of the previous studies on retroperitoneal TLH were small case series or retrospective comparative studies with conventional TLH. Therefore, the investigators conducted this randomized trial to investigate the role of retroperitoneal TLH in enlarge uterus.

ELIGIBILITY:
Inclusion Criteria:

* absence of pregnancy at the time of presentation
* uterine volume between 12 and 18 weeks of gestation by pelvic examination
* appropriate medical status for laparoscopic surgery (American Society of Anesthesiologists Physical Status classification 1 or 2)

Exclusion Criteria:

* any suggestion of malignant uterine or adnexal diseases
* any major medical comorbidities or psychiatric illnesses, which could affect follow-up and/or compliance
* an inability to understand and provide written informed consent.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Operative blood loss | Operation day
  Operative blood loss was calculated by the anesthesiology unit as the difference between the total amount of suction and irrigation plus the difference between the total gauze weight before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Study Chair — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No